CLINICAL TRIAL: NCT05429918
Title: A Multicenter Prospective Observational Study to Evaluate the Safety and Efficacy of Ibrutinib Combined With R-CHOP/R-DHAP in Newly Diagnosed Mantle Cell Lymphoma Patients Who Aged ≤65 Years
Brief Title: Ibrutinib Combined With R-CHOP/R-DHAP in Newly Diagnosed Mantle Cell Lymphoma Patients Who Aged ≤65 Years
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Collaborators: The Second Affiliated Hospital of Dalian Medical University (Other); Peking University First Hospital (Other); Beijing Hospital (Other Government); Beijing Tsinghua Changgeng Hospital (Other); China-Japan Friendship Hospital (Other); Chinese PLA General Hospital (Other); First Affiliated Hospital of Harbin Medical University (Other); Baotou Cancer Hospital (Other); Beijing Shijitan Hospital, Capital Medical University (Other); Shanxi Province Cancer Hospital (Other); Beijing Naval General Hospital (Other); First Hospital of China Medical University (Other); Jilin Provincial Tumor Hospital (Other); Shengjing Hospital (Other); 307 Hospital of PLA (Other); Peking Union Medical College Hospital (Other); Harbin Medical University (Other); Beijing Tongren Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2021028
Record Dates: First submitted 2021-07-08; First posted 2022-06-23 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2022-06

CONDITIONS: Mantle Cell Lymphoma
Keywords: MCL; ibrutinib; aged ≤65 years
MeSH Terms: conditions — Lymphoma, Mantle-Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The purpose of the study is to better and systematically collect clinical data on the treatment of ibrutinib combined with R-CHOP/DHAP regimen for more scientific and accurate evaluation, our center has carried out the R-CHOP/R-DHAP alternative regimen combined with ibrutinib at age ≤ An observational clinical study on the safety and effectiveness of 65-year-old mantle cell lymphoma. Through this study, young mantle cell lymphomas in the Chinese population can be collected. Ibrutinib combined with R-CHOP/R-DHAP is used in the initial treatment. 2 and 6 cycles of ORR were used to evaluate survival indicators, and collect adverse reactions during treatment and recurrence rate after treatment.

DETAILED DESCRIPTION:
Mantle cell lymphoma (MCL) is a B-cell lymphoma with unique histomorphology、immunophenotype and cytogenetic characteristics, accounting for 6% to 8% of non-hodgkin's lymphoma, occurs in older men, median age 68 years old, male: female is about 2 to 4:1, 80% of patients during the diagnosis is in progress, both indolent and aggressive lymphoma inert lymphoma incurable characteristic. The main clinical manifestations were lymph node, hepatosplenomegaly. Extranodal involvement is common, and the commonly involved sites include bone marrow, gastrointestinal tract, and Waldeyer'sring [1], t (11; 14) (q13; q32) Excessive expression in the Cyclin D1 nucleus caused by abnormalities is characteristic of MCL.In recent years, although the application of new drugs has made a lot of progress in the treatment of mantle cell lymphoma, the overall efficacy is not good, the vast majority of patients relapse after treatment, the median survival of 3-5 years, the lack of standard treatment regimens[2.3]. Blast-cell type and high-risk mantle cell lymphoma account for 10-15%, with higher clinical invasiveness and poorer prognosis.Mantle cell lymphoma responds to combination therapy, but easy to relapse is still a difficult point in clinical treatment. Rituximab combined with chemotherapy can increase the effective rate of treatment and prolong the median survival time, but it does not significantly improve the overall survival rate[4] . For young patients with good general conditions, it is currently believed that the intensive treatment of high-dose cytarabine should be selected first as induction therapy, and then sequential autologous hematopoietic stem cell transplantation should be used as consolidation therapy. Romaguera et al. [4] reported the efficacy of R-hyperCVAD A/B regimen in 97 newly-treated MCL patients. The results showed that the 3-year FFS and OS of MCL patients younger than 65 were 73% and 82%, respectively, but the bone marrow suppression effect of this program is obvious, and the risk of infection is increased. It is not recommended for elderly patients with poor general conditions[6,7] . The results of the GELA study on the application of R-CHOP/R-DHAP sequential autologous stem cell transplantation in newly-treated MCL showed that the median EFS was 83.9 months, the median OS did not reach, and the 5-year OS was 75%, and no treatment-related mortality occurred. , Indicating that the combination chemotherapy regimen based on rituximab and cytarabine is a safe and effective treatment regimen for MCL[7] . In the European Mantle Cell Lymphoma Collaborative Group's randomized, open-ended, multicenter phase III clinical study on the application of high-dose cytarabine in initial mantle cell lymphoma, R -CHOP or R-CHOP/R-DHAP program sequential auto-HSCT curative effect compared with the control group, although the side effects of bone marrow suppression increased, but the disease progression time of the treatment group containing high-dose cytarabine was significantly prolonged, 9.1 vs 3.9 years (P=0.038). A number of studies believe that rituximab combined with high-dose cytarabine chemotherapy and sequential autologous hematopoietic stem cell transplantation is the first-line treatment for patients with MCL aged ≤65 years[9，10] . Despite the existence of the above-mentioned first-line and data programs, 60% of patients with mantle cell lymphoma in clinic have disease recurrence after first-line treatment. Therefore, how to improve the depth of remission and reduce disease recurrence in newly treated mantle cell lymphoma patients has become the treatment of mantle cell lymphoma. Important goals.Ibrutinib, as a BTK inhibitor, has shown significant efficacy in the treatment of mantle cell lymphoma, and has become an important choice in the treatment of mantle cell lymphoma[11] .The PCYC1104 clinical study showed that ibrutinib monotherapy was used to treat recurrent and refractory mantle cell lymphoma with a median follow-up of 15.3 months, with a CR21%, PR47%, ORR68%, and a median PFS13.9 months[12,13];Another randomized, open, multi-center phase III trial comparing ibrutinib to Temsirolimus monotherapy in relapsed and refractory mantle cell lymphoma showed a statistically significant difference in CR18.7%,PR53.2%, ORR72%and median PFS15.6 months compared with sirolimus monotherapy[14]. Based on these studies, ibrutinib is now an important treatment option for relapsed and refractory mantle cell lymphoma recommended by various guidelines.The significant efficacy of ibrutinib in the treatment of mantle cell lymphoma has been studied both at home and abroad. Ibrutinib is used for the treatment of patients with mantle cell lymphoma at the initial treatment, and combined treatment with ibrutinib can achieve deep complete remission and reduce disease recurrence. In 2019, MD Anderson of the United States carried out a clinical study of ibrutinib combined with rituximab in the treatment of initial mantle cell lymphoma. 50 patients with newly treated mantle cell lymphoma were included. After remission was induced by the IR regimen, the subsequent combined hyperCAVD A/B regimen was alternately consolidated. For 4 cycles, the above study showed that ORR was 100%, 3-year PFS 88%, 3-year OS 100%, and there was no significant difference in PFS between the ki67 proliferation high-risk group and the low-risk group. The above study was ibrutinib combined Treatment provides a basis for treatment in newly-treated mantle cell lymphoma, and has become an important treatment option for newly-treated mantle cell lymphoma.The retrospective analysis of 256 cases of Chinese patients with mantle cell lymphoma showed that the survival rate of Chinese patients with mantle cell lymphoma after initial treatment was 40.9%, Orrin 81.6%, 5-year PFS 51.2% and 5-year OS 58.4%, which were significantly lower than that of foreign patients with mantle cell lymphoma. Survival of patients with mantle cell lymphoma in China; At the same time, 56.8% of patients relapsed after the disease was remission, and the overall treatment effect was not good after the relapse. Therefore, the initial treatment of mantle cell lymphoma patients for the Chinese population needs to be further optimized. As the longest time-to-market BTK inhibitor in the clinic, Ibrutinib has been widely used in the clinical treatment of mantle cell lymphoma and is also included in the scope of medical insurance reimbursement. As the longest time-to-market BTK inhibitor in the clinic, Ibrutinib has been widely used in the clinical treatment of mantle cell lymphoma and is also included in the scope of medical insurance reimbursement. In clinical treatment, Ibrutinib combined with R-CHOP/DHAP regimen has been used for treatment, which has shown a good complete remission rate, and at the same time the safety is tolerable. In order to better and systematically collect clinical data on the treatment of ibrutinib combined with R-CHOP/DHAP regimen for more scientific and accurate evaluation, our center has carried out the R-CHOP/R-DHAP alternative regimen combined with ibrutinib at age ≤ An observational clinical study on the safety and effectiveness of 65-year-old mantle cell lymphoma. Through this study, young mantle cell lymphomas in the Chinese population can be collected. Ibrutinib combined with R-CHOP/R-DHAP is used in the initial treatment. 2 and 6 cycles of ORR were used to evaluate survival indicators, and collect adverse reactions during treatment and recurrence rate after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. age 18-65 years old;
2. The pathological biopsy was consistent with mantle cell lymphoma;
3. Measurable lesions on cross-sectional imaging recorded by diagnostic imaging (computed tomography [CT] or magnetic resonance imaging [MRI]) (defined as the presence of at least one two-dimensional measurable lesion with a maximum cross-sectional diameter (GTD) ≥1.5 cm, regardless of the short axis diameter);
4. The physical status of the Eastern United States Cooperative Oncology Group (ECOG) ≤2 points;
5. Full liver function: upper limit of bilirubin≤3×normal value (ULN);Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤5×ULN; Alkaline phosphatase (ALP) ≤5×ULN; Serum creatinine ≤1.5×ULN, or creatinine clearance rate calculated according to Cockcroft-Gault formula ≥35mL/min;
6. Voluntary participation, willingness to provide the above treatment data, signed and dated informed consent -

Exclusion Criteria:

1. Other clinical trials have been included;
2. Immunosuppressive therapy is being used for other diseases;
3. Lymphoma has been treated with other regimens before entry;
4. Complicated with other malignant tumors;
5. Those who are judged by the investigator to be unsuitable to participate in this study;
6. Serious mental or neurological disorder that affects informed consent and/or the presentation or observation of adverse reactions;
7. Patients who could not be followed up

Exit (drop-off) criteria :

1. Subject requires to quit;
2. Serious adverse events occurred during the trial, so it is inappropriate to continue the clinical trial;
3. If the disease progresses during the study, it is inappropriate to continue using the experimental drug and/or cannot continue the study protocol;
4. Incomplete research data records;
5. Patients could not be followed up.Withdrawal cases should be retained for future reference and transferred from the last record to the final record for ITT analysis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 60 patients with primary mantle cell lymphoma
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-12-30 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
the overall response (complete response + partial response) | From the date of first study drug administration until the end of Cycle 2 (each cycle is 28 days)
  Objective response rate，sum of complete response rate and partial response rate of ibrutinib combination therapy in initial treatment of MCL
the overall response (complete response + partial response) | From the date of first study drug administration until the end of Cycle 6 (each cycle is 28 days)
  Objective response rate，sum of complete response rate and partial response rate of ibrutinib combination therapy in initial treatment of MCL

SECONDARY OUTCOMES:
Progression-free survival (PFS),OS,CR,DOR | 2years
  Efficacy and survival of ibrutinib combination therapy in primary MCL, including: PFS,OS,CR,DOR
Incidence and severity of adverse events(AE) | 2 years
  Incidence of toxicity, defined as grade 3 or higher non-hematologic toxicity, grade 3 neutropenia, grade 4 hematologic toxicity, inability to administer full schedule and dose, or inability to receive treatment day 1 of course 2
The recurrence rate of MCL after initial treatment with ibrutinib | 2years
  The recurrence rate of MCL after initial treatment with ibrutinib
Minimal residual disease negative (MRD-) rate of patients combination therapy | 1year and 2years
  MRD- rate will be estimated as the percentage of patients who achieved MRD-(ctDNA from Peripheral blood determined by NGS).

CONTACTS AND LOCATIONS:
Overall Officials: Hongmei Jing, Professor, Study Chair — Peking University Third Hospital
Locations (1):
- Hongmei Third Jing, Beijing, Beijing Municipality, China